CLINICAL TRIAL: NCT01455207
Title: From Uncomplicated Alcoholism to Korsakoff's Syndrome: Clinical, Genetic, Neuropsychological and Brain Examinations
Brief Title: From Uncomplicated Alcoholism to Korsakoff's Syndrome
Acronym: ALCOBRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A00495-36; 11-050
Record Dates: First submitted 2011-10-18; First posted 2011-10-19 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Alcoholism; Alcohol Amnestic Disorder
Keywords: Magnetic Resonance Imaging; Positon Emission Tomography; Behavior
MeSH Terms: conditions — Alcoholism; Alcohol Amnestic Disorder; Behavior | interventions — Neuropsychological Tests; Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- alcoholic patients (Other)
  Interventions: Behavioral: Neuropsychological testing; Biological: blood draw; Genetic: genetic testing; Other: Brain imaging examination
- korsakoff patients (Other)
  Interventions: Behavioral: Neuropsychological testing; Biological: blood draw; Genetic: genetic testing; Other: Brain imaging examination
- healthy controls (Other)
  Interventions: Behavioral: Neuropsychological testing; Biological: blood draw; Genetic: genetic testing; Other: Brain imaging examination

INTERVENTIONS:
Behavioral: Neuropsychological testing — assessment of memory, executive functions and ataxia
Biological: blood draw — hepatic markers, red blood markers and vitamin markers
Genetic: genetic testing — genes coding for thiamine enzymes (α-ketoglutarate dehydrogenase complex, transketolase et pyruvate dehydrogenase)
Other: Brain imaging examination — MRI, DTI and PET examinations

SUMMARY:
This research project aims to identify factors that contribute to the heterogeneity observed in neuroradiological and neuropsychological signs of chronic alcoholism. The investigators overarching hypothesis is that the heterogeneity of alcoholic consequences on brain structure and metabolism, and cognition is mainly related to individual differences in pattern of alcohol use, gene pool, nutritional status and history of withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Completed at least 8 years of education (primary school equivalent)
* Age-normal corrected hearing and visual acuity

Exclusion Criteria:

* documented loss of consciousness of over 30 minutes, documented compound skull fracture, or clear neurological sequelae of head trauma
* history of medical or neurological illness or trauma potentially affecting the CNS, e.g., stroke, multiple sclerosis, epilepsy, psychosurgery, insulin coma.
* active tuberculosis or history of or any malignancy requiring chemotherapy
* history of schizophrenia or bipolar disorder
* metal implantation (e.g., pacemakers) or other factors that preclude MRI scanning for subjects selected for the neuroimaging examination
* meet DSM-IV criteria for current (past 3 months) other Substance Abuse
* met DSM-IV criteria for other Substance Dependence
* Have used other substances more than 5 times in the past month

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of brain dysfunctioning measured by neuropsychological testing and brain examination(MRI and PET) | one year

SECONDARY OUTCOMES:
treatment outcomes (sobriety or relapse) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France